CLINICAL TRIAL: NCT01488799
Title: Adding Motivational Interviewing to Cognitive Behavioural Therapy for Severe Generalized Anxiety Disorder
Brief Title: Motivational Interviewing and Cognitive Behavioural Therapy for Generalized Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Collaborators: Toronto Metropolitan University (Other); University of Massachusetts, Amherst (Other)
Responsible Party: Principal Investigator, Henny Westra, Clinical Psychologist, Associate Professor (York University), York University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOP114909
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Anxiety Disorders; Generalized Anxiety Disorder
Keywords: Anxiety; Generalized Anxiety Disorder; Motivational Interviewing; Cognitive Behavioural Therapy; Psychotherapy
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder | interventions — Motivational Interviewing; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MI-CBT (Active Comparator)
  Interventions: Behavioral: Motivational Interviewing and Cognitive Behavioural Therapy
- CBT alone (Active Comparator)
  Interventions: Behavioral: Motivational Interviewing and Cognitive Behavioural Therapy

INTERVENTIONS:
Behavioral: Motivational Interviewing and Cognitive Behavioural Therapy — Participants with a diagnosis of severe Generalized Anxiety Disorder will be randomly assigned to receive either 4 weekly sessions of MI followed by 11 weekly sessions of CBT (MI-CBT arm) or 15 weekly sessions of CBT (CBT alone arm). Both groups will also receive 2 follow-up CBT treatment sessions at 1 and 3 months post-treatment. In order to increase generalizability to clinical practice, in the CBT phase for the MI-CBT arm, therapists will shift to MI in the presence of empirically derived markers of resistance and shift back to CBT when resistance has diminished. In the CBT alone arm therapists will respond to resistance using manualized recommendations derived from leading CBT theorists for the management of resistance.
  Other Names: Motivational Interviewing; Cognitive Behavioral Therapy

SUMMARY:
The current study examines whether change-readiness, and consequently treatment outcome, can be enhanced in Cognitive Behavioral Therapy (CBT) for severe Generalized Anxiety Disorder (GAD) by adding a brief course of Motivational Interviewing (MI adapted for anxiety, Westra & Dozois, 2003) before and during CBT when motivation wanes. 106 individuals with severe GAD will be randomly assigned to receive an equal number of sessions of either MI and CBT (MI-CBT arm) or CBT alone (CBT alone arm). It is expected that the MI-CBT arm relative to the CBT alone arm will show lower levels of resistance in CBT, higher levels of homework compliance and therapeutic alliance, better moment-to-moment interpersonal process, and consequently superior outcomes - both post-treatment and at 6 and 12 month follow-ups.

DETAILED DESCRIPTION:
The proposed study builds on the findings of the clinical trial by Westra, Arkowitz and Dozois (2009), and aims to: (1) provide a powerful test of the value of adding MI to CBT for high severity GAD (as pilot data has indicated that individuals with severe GAD may preferentially benefit from the addition of MI to CBT), (2) employ treatment procedures generalizable to clinical practice, and (3) examine the mechanisms underlying any additive treatment benefit. 106 individuals with a principal diagnosis of GAD and of high worry severity will be randomly assigned to receive either 4 sessions of MI followed by 11 sessions of CBT (MI-CBT arm) or 15 sessions of CBT (CBT alone arm). Both groups will also receive 2 follow-up CBT treatment sessions at 1 and 3 months post-treatment. Each therapist will deliver all treatment components, treatments will appear seamless to clients, and therapists will be nested within treatment group to control for allegiance effects and avoid cross-contamination of the therapies. In order to increase generalizability to clinical practice, in the CBT phase for the MI-CBT arm, therapists will shift to MI in the presence of empirically derived markers of resistance and shift back to CBT when resistance has diminished. In the CBT alone arm therapists will respond to resistance using manualized recommendations derived from leading CBT theorists for the management of resistance. Anxiety and related symptoms, motivation, and treatment engagement will be assessed at various points during treatment, and at 6 and 12 months post-treatment. A multi-method approach to assessment will be used, including self-report, clinician-report, clinician-administered, observer-rated, and interview-based measures. Importantly, we will include not only traditional outcome measures, but also process measures (e.g., observer-coded interpersonal behavior, interview-based derivation of client experiences) to investigate possible mechanisms underlying any additive treatment benefit. In addition, all therapy sessions will be videotaped and assessed by independent raters for protocol adherence.

The specific hypotheses are as followed:

Hypothesis 1: Worry, Anxiety, & Related Symptoms. The MI-CBT arm will show greater reductions in worry, anxiety, and related symptoms (depression, disability, maladaptive beliefs about worry, life satisfaction) and a greater percentage of treatment responders (using clinical significance criteria) across the treatment period and at follow-up (FU), compared to the CBT alone arm.

Hypothesis 2: Motivation and Resistance. Over the course of early treatment (i.e., sessions 1 to 4), the MI-CBT arm will demonstrate greater increases in motivation compared to the CBT alone arm. In addition, the MI-CBT arm will exhibit lower in-session resistance during early (sessions 5 & 7), middle (sessions 10 & 12), and late (sessions 15 & 17) phases of treatment.

Hypothesis 3: Homework Compliance. The MI-CBT arm will show greater client- and therapist-rated homework compliance throughout CBT treatment compared to the CBT alone arm.

Hypothesis 4a: Interpersonal Processes between Clients and Therapists. Compared to CBT alone clients, MI-CBT clients and therapists will report higher working alliance quality during both the initial MI sessions and subsequent phases of CBT. Furthermore, moment-to-moment interpersonal processes between client and therapist during early, middle, and late treatment are expected to be characterized by more adaptive processes (e.g., higher affiliation and less hostility) in the MI-CBT vs. CBT alone arms.

Hypothesis 4b. Interpersonal Processes During Resistance. During episodes of client resistance (identified with resistance coding), therapist and client exchanges in MI-CBT are expected to be characterized by more adaptive processes (i.e., higher affiliation, less hostility, and greater client autonomy-preservation) compared to CBT alone. Further, when a small subset of clients (5 per treatment group) are interviewed about their experiences of resistance episodes, we expect client accounts in the MI-CBT arm to be characterized more positively (e.g., more supportive of client autonomy, more conducive to increased engagement vs. disengagement with treatment) compared to CBT alone.

Hypothesis 5: Mediation of Therapeutic Outcomes. We expect that increased motivation and reduced resistance in MI-CBT, compared to CBT alone, will lead to higher levels of engagement in the CBT (better homework compliance and therapeutic alliance), which will result in greater worry reduction.

ELIGIBILITY:
Inclusion Criteria:

* Between 16 & 65 years of age
* Proficient use of English
* A principle diagnosis of Generalized Anxiety Disorder (GAD)
* Severe GAD (as measured by clinician severity ratings and PSWQ)
* Willingness to either remain on stable dosage of psychotropic medication or remain unmedicated throughout their involvement in the clinical trial

Exclusion Criteria:

* Current of history of psychotic spectrum disorder or bipolar mood disorder
* Cognitive impairment such as neurodegenerative illness or head injury
* Current substance abuse and or dependance
* Concurrent psychotherapy, either individual or group.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2012-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Penn State Worry Questionnaire (PSWQ) | up to 4 years
  The Penn State Worry Questionnaire (PSWQ; Meyer et al., 1990) is a widely used measure of worry in GAD treatment outcome studies. It is a 16-item scale assessing trait worry. The PSWQ has been found to possess high internal consistency and temporal stability, as well as good convergent and discriminant validity. It also differentiates individuals with GAD from those with other anxiety disorders (Brown et al., 1992).

SECONDARY OUTCOMES:
Satisfaction with Life Scale (SWLS) | up to 4 years
  The Satisfaction with Life Scale (SWLS; Diener et al., 1985)is a 5-item scale that is a widely used as a measure of life satisfaction with high internal validity, temporal stability, and sensitivity to change, as well as good convergent and divergent validity.
Inventory of Interpersonal Problems (IIP) | up to 4 years
  The Inventory of Interpersonal Problems (IIP; Horowitz, Rosenberg, Baer, Ureño, & Villaseñor, 1988), scale has been shown to discriminate among different categories of personality disorders and reliably tap into three dimensions of the the interpersonal relational field (Gude, Moum, Kaldestad, & Friis, 2000).
Depression Anxiety Stress Scale (DASS) | up to 4 years
  The Depression Anxiety Stress Scale (DASS; Lovibond & Lovibond, 1995) is a set of three self-report scales designed to define, measure and understand depression, anxiety and stress. Each scale contains 14 items, for a total of 42 items, and each scale is divided into sub-scales of 2-5 items based on content. The DASS shows strong consistent reliability in distinguishing between features of depression, anxiety and stress (Antony, Bieling, Cox, Enns, Murray & Swinson, 1998).

CONTACTS AND LOCATIONS:
Overall Officials: Henny A Westra, Ph.D., Principal Investigator — York University; Martin M Antony, Ph.D., Principal Investigator — Toronto Metropolitan University; Michael J Constantino, Ph.D., Principal Investigator — University of Massachusetts, Worcester
Locations (2):
- Canada (2):
  - York University, Toronto, Ontario
  - Ryerson University, Toronto, Ontario